CLINICAL TRIAL: NCT02523625
Title: Can we Use Ultrasound in the Diagnosis and Monitoring of Patients With Giant Cell Arteritis?
Brief Title: Giant Cell Arteritis: Improving Use of Ultrasound Evaluation
Acronym: GAULT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oxford (Other)
Collaborators: University of Lisbon (Other)
Responsible Party: Sponsor
Other Study IDs: 9776
Record Dates: First submitted 2015-08-04; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Giant Cell Arteritis
Keywords: Ultrasound
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy volunteers: Age and gender matched to patient groups to undergo ultrasound of temporal and axillary arteries
  Interventions: Device: Ultrasound of temporal and axillary arteries
- Patients with headache: Patients with new headache not due to GCA to undergo ultrasound of temporal and axillary arteries
  Interventions: Device: Ultrasound of temporal and axillary arteries
- Patients with GCA (new): Patients with new diagnosis of GCA to undergo ultrasound of temporal and axillary arteries
  Interventions: Device: Ultrasound of temporal and axillary arteries
- Patients with GCA (flare): Patients with apparent flare of GCA to undergo ultrasound of temporal and axillary arteries
  Interventions: Device: Ultrasound of temporal and axillary arteries

INTERVENTIONS:
Device: Ultrasound of temporal and axillary arteries — Each patient will have a clinical assessment and ultrasound examination of both temporal and axillary arteries

SUMMARY:
Giant cell arteritis (GCA) is an inflammatory disease causing new, unaccustomed headache in the elderly and which can lead to blindness in 20-30% of untreated cases. The study group have previously shown that ultrasound is a viable non-invasive alternative to temporal artery biopsy in diagnosing GCA. However, there is significant variation in ultrasound assessment (measuring a dark "halo" around the abnormal blood vessels) between sonographers in different centres, requiring a labour intensive and time consuming training programme. The study group propose to standardise the training programme, and use ultrasound and clinical evaluation to define changes occurring over time and with treatment in patients with a diagnosis of GCA made based on ultrasound changes alone. The study group will explore the use of algorithms to automate or semi-automate image interpretation.

DETAILED DESCRIPTION:
Objectives and Project Plan:

* Project Purpose:

The purpose of the project is to develop the technology to reliably acquire and analyse ultrasound images through the use of a training programme which are comparable to those from scanning by an expert sonographer in the diagnosis (i.e. as a diagnostic tool) and monitoring of patients with GCA following treatment (i.e. as a response indicator), and patient stratification according to initial or early scan changes to determine the most appropriate treatment (i.e. as a prognostic tool).

* End Point:

The end point will be the production of an effective training programme which can be used to obtain reproducible accurate ultrasound images of the temporal artery which can be automatically analysed and used in real time in the management of patients with suspected or confirmed giant cell arteritis.

* Milestones:

The project is in 3 phases. In phase 1 (0-12 months) the study group will create a bank of images for training from healthy volunteers and patients with GCA; in phase 2 (13-18 months) the study group will test the programme on sonographers assessing patients with GCA; in phase 3 (19-42 months) the study group will acquire serial images, clinical data, serum and plasma from cohorts of patients with newly diagnosed and flaring GCA so that they can analyse and develop new software algorithms. The study group can use images already acquired from a previous diagnostic study in GCA, and test the algorithms on the new cohorts..

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer or
* Patient with a suspected diagnosis of GCA but found not to have GCA
* Recent diagnosis of GCA within 1 month or
* Suspected flare of GCA within one month
* Ability to provide written informed consent

Exclusion Criteria:

* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or diagnosed giant cell arteritis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Size of halo detected (mm) on ultrasound of temporal arteries | 24 months
  The study group will compare computer algorithms to analyse the halo size from video images of ultrasound scans with observer defined measures of halo size (mm) from healthy volunteers, patients with headache but not due to GCA, patients with newly diagnosed GCA and in patients with GCA who are followed serially and re-imaged over time in response to therapy. The study group will test the value of algorithms incorporating clinical and serological data together with the imaging findings to determine their added effect on the sensitivity and specificity of ultrasound for diagnosis and monitoring of GCA. Halo size varies from 0 (undetectable) to greater than 1mm. Cut-off values for abnormal values have not been formally established or published yet.

SECONDARY OUTCOMES:
Circulating serum Vascular Endothelial Growth Factor (VEGF) levels | 24 months
  The study group will measure VEGF levels in serum taken from age matched controls presenting with headache, patients with newly diagnosed GCA and patients with established GCA undergoing a flare, to determine the value of VEGF in predicting diagnosis, response to therapy, flare or prognosis in GCA.
Circulating serum Pentraxin 3 levels | 24 months
  The study group will measure pentraxin 3 levels in serum taken from age matched controls presenting with headache, patients with newly diagnosed GCA and patients with established GCA undergoing a flare, to determine the value of pentraxin 3 in predicting diagnosis, response to therapy, flare or prognosis in GCA.

CONTACTS AND LOCATIONS:
Overall Officials: Raashid A Luqmani, DM FRCP, Principal Investigator — University of Oxford

REFERENCES:
- [Result] Ponte C, Rodrigues AF, O'Neill L, Luqmani RA. Giant cell arteritis: Current treatment and management. World J Clin Cases. 2015 Jun 16;3(6):484-94. doi: 10.12998/wjcc.v3.i6.484. PMID 26090367
- [Result] Diamantopoulos AP, Myklebust G. Long-term inflammation in the temporal artery of a giant cell arteritis patient as detected by ultrasound. Ther Adv Musculoskelet Dis. 2014 Jun;6(3):102-3. doi: 10.1177/1759720X14521109. No abstract available. PMID 24891881
- [Result] Schmidt WA. Ultrasound in vasculitis. Clin Exp Rheumatol. 2014 Jan-Feb;32(1 Suppl 80):S71-7. Epub 2014 Feb 17. PMID 24529335
- [Result] Diamantopoulos AP, Haugeberg G, Hetland H, Soldal DM, Bie R, Myklebust G. Diagnostic value of color Doppler ultrasonography of temporal arteries and large vessels in giant cell arteritis: a consecutive case series. Arthritis Care Res (Hoboken). 2014 Jan;66(1):113-9. doi: 10.1002/acr.22178. PMID 24106211
- [Result] Muratore F, Boiardi L, Restuccia G, Macchioni P, Pazzola G, Nicolini A, Germano G, Possemato N, Cavazza A, Cavuto S, Cimino L, Pipitone N, Catanoso M, Addimanda O, Salvarani C. Comparison between colour duplex sonography findings and different histological patterns of temporal artery. Rheumatology (Oxford). 2013 Dec;52(12):2268-74. doi: 10.1093/rheumatology/ket258. Epub 2013 Sep 17. PMID 24046471
- [Result] Habib HM, Essa AA, Hassan AA. Color duplex ultrasonography of temporal arteries: role in diagnosis and follow-up of suspected cases of temporal arteritis. Clin Rheumatol. 2012 Feb;31(2):231-7. doi: 10.1007/s10067-011-1808-0. Epub 2011 Jul 9. PMID 21743987